CLINICAL TRIAL: NCT04405063
Title: A Prospective, Multicenter, Sponsor Initiated, Randomized Controlled Trials to Evaluate the Safety and Efficacy of Genoss® DCB Compared to Sequent® Please in Korean Patients With Coronary Artery In-stent Restenosis (ISR)
Brief Title: Compare the Safety and Efficacy of Genoss® DCB and SeQuent® Please in Korean Patients With Coronary In-stent Restenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genoss Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP-DS1001
Record Dates: First submitted 2020-05-18; First posted 2020-05-28 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease
Keywords: In-Stent Restenosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genoss® DCB (Experimental): Paclitaxel Coated PTCA Balloon Catheter
  Interventions: Device: Paclitaxel Coated PTCA Balloon Catheter
- SeQuent® Please (Active Comparator): Paclitaxel Coated PTCA Balloon Catheter
  Interventions: Device: Paclitaxel Coated PTCA Balloon Catheter

INTERVENTIONS:
Device: Paclitaxel Coated PTCA Balloon Catheter — Drug coated balloon

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Paclitaxel-coated balloon (Genoss® DCB) by demonstrating non-inferiority to in-segment late lumen loss at 6 months after the procedure in patients with in-stent restenosis (ISR) compared with a product of the same category (Sequent® Please)

DETAILED DESCRIPTION:
In a randomized controlled trials to compare with the same-category medical device (Sequent® Please), 82 patients with in-stent restenosis (ISR) were recruited from a total of 7 institutions, and the enrolled subjects were 1: 1 through randomization. The ratio was assigned to the test group and the control group, and each of the test or control devices was assigned to receive the procedure.

Drug release "stents" for PCI usually follow 9 months or 12 months, but the medical device for this clinical trial has a drug coated "balloon catheter" and the mechanism of action is different from the stent and the duration of follow up was set to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 years old
* Patients with significant coronary artery stenosis including left main coronary lesion (> 50% diameter stenosis on coronary angiography)
* Patients with stable angina pectoris, or unstable angina pectoris, and asymptomatic myocardial ischemia
* Patients suitable to receive coronary revascularization of any type
* Restenosis Mehran type I-III after stent implantation for the first time
* Patients with In-stent restenosis after 90 days of the stent implantation, and the degree of restenosis corresponds to Mehran type I-Ⅲ.
* Diameter of the stent with restenosis should be 2.0-4.0mm (included). Length of the stenosis lesion should be no more than 40mm
* In case of voluntarily deciding to participate in this clinical trial by signing the informed consent form

Exclusion Criteria:

* Patients with Infarct related artery (IRA) lesions among patients with acute myocardial infarction
* Patients have restenosis lesions with thrombosis
* Patients with a history of cardiogenic shock
* Patients with total occlusion indicating TIMI 0 blood flow at the target lesion (Mehran type IV stenosis)
* Patients with graft vessel lesion
* Patients who are contraindicated in aspirin, heparin, clopidogrel, ticlopidine, and paclitaxel
* Patients with renal insufficiency (eGFR<30mL/min)
* Pregnant or lactating women
* The patients have a life expectancy of less than 12 months
* Patients who had reduced immunity or clinically significant abnormalities in the laboratory tests (hematological, serum biochemical, and urine tests) performed at the time of screening
* Patients who had clinically significant disorders in cardiovascular system, digestive system, respiratory system, endocrine system, and central nervous system, or mental illness that significantly affects this study
* Patients who are unsuitable for the study according to the investigator judges

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
In-segment late lumen loss after percutaneous coronary intervention in patients with ISR | Follow-up angiography at 6 months after procedure
  In-segment late lumen loss between test group(Genoss DCB) and control group(Sequent Please) evaluated by quantitiative coronary analysis in patients with ISR

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jun EJ, Shin ES, Yuan SL, Bhak Y, Garg S, Kang WC, Kim JS, Kim JH, Bae JW, Rha SW, Chae IH. Comparison of 2 Different Paclitaxel-Coated Balloons in Coronary In-Stent Restenosis: A Randomized Controlled Trial. JACC Asia. 2022 Mar 1;2(2):170-179. doi: 10.1016/j.jacasi.2021.11.015. eCollection 2022 Apr. PMID 36339121